CLINICAL TRIAL: NCT03047135
Title: Phase II Study of Olaparib in Men With High-Risk Biochemically-Recurrent Prostate Cancer Following Radical Prostatectomy, With Integrated Biomarker Analysis
Brief Title: Olaparib in Men With High-Risk Biochemically-Recurrent Prostate Cancer Following Radical Prostatectomy, With Integrated Biomarker Analysis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J16163; IRB00114635 (Other: JHM IRB)
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Results first posted 2024-07-03 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Prostate
Keywords: high-risk biochemically-recurrent
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olaparib 300 mg BID (Experimental): Patients will be administered olaparib orally twice daily at 300mg bid continually. Two 150mg of olaparib tablets should be taken twice daily, approximately 12 hours apart with one glass of water.
  Interventions: Drug: Olaparib

INTERVENTIONS:
Drug: Olaparib — Olaparib will be dispensed to patients on Day 1 and every 28 days thereafter until the patient completes the study, withdraws from the study or closure of the study.

SUMMARY:
Olaparib has demonstrated preliminary efficacy in metastatic castration-resistant prostate cancer. In a trial of 49 evaluable patients treated with olaparib, 11 / 49 experienced a PSA response, and every patient with a radiographic response also had a PSA5 response.

Ten of 11 responders had mutations in DNA repair genes. While PARP inhibition is showing promise in these initial studies, reserving its use for end-stage patients may not be the optimal timing for olaparib therapy in some patients. In addition, PARP enzymes function in roles beyond DNA repair, and specifically for prostate cancer are involved transcriptional regulation of the androgen receptor. PARP inhibition has not been tested in earlier disease states for prostate cancer.

DETAILED DESCRIPTION:
The proposed study is an open-label single-arm phase II trial.

Eligible patients are those with non-metastatic biochemically-recurrent prostate cancer and a PSADT of ≤6 months and a minimum PSA of 1.0.

After enrollment, patients will be treated with olaparib at the established dose of 300mg tablets by mouth twice daily. Patients will be followed monthly with clinic visits, safety labs (including CBC w/diff, Comp), PSA, and toxicity assessments. Treatment [with a minimum drug exposure of 12 weeks] will be continued until PSA doubling from study entry (confirmed with another measurement at least 4 weeks later), development of radiographic metastatic disease, or toxicity requiring drug cessation. CT scans and NM bone scans will be performed every 6 months for patients remaining on olaparib treatment.

This study will enroll up to 50 subjects. The study design will employ a stepwise adaptive statistical plan, derived in part from Biankin et al, Nature 2015 Oct 15;526(7573):361-70. The design is adapted from a multi-stage design, with interim stopping rules to determine futility or need for enrichment of the study population.

The study will initiate with a two-stage design in an unselected population. The assumptions for the trial of the unselected population are: null hypothesis of 0.1 PSA response rate and alternative hypothesis of 0.3 for the unselected population. The first stage is 20 subjects. If ≤2 subjects responds in the first stage, then unselected population study is halted for futility and an assessment of DNA mutations present in the initial cohort will be undertaken. If less than 3 subjects with a known/suspected deleterious mutation in the following genes (ATM, BARD1, BRCA1, BRCA2, BRIP1, CDK12, CHEK1, CHEK2, FANCL, PALB2, PPP2R2A, RAD51B, RAD51C, RAD51D, or other DNA repair genes) have been accrued in the first stage, then the trial will proceed with enrichment. If 3 or more subjects with known/suspected deleterious mutation in the genes of interest have been accrued, then the trial will proceed with enrichment, as long as the response rate in that subset of subjects is ≥20%. In the case that 3 or more subjects have been accrued, yet the response rate in that subset is <20%, then the trial is halted for futility.

However, if ≥3 subjects among the first 20 respond, then additional 10 unselected subjects are accrued. If ≥6 subjects respond out of 30 in the unselected population after the second stage, then the null hypothesis is rejected in the unselected population and broad efficacy will be concluded.

The trial proceeds to complete accrual of 50 subjects in order to better estimate PSA response rate and strengthen data for correlative studies. If <6 respond, then the null hypothesis is not rejected. Again, if less than 3 subjects with a known/suspected deleterious mutation in the following genes (ATM, BARD1, BRCA1, BRCA2, BRIP1, CDK12, CHEK1, CHEK2, FANCL, PALB2, PPP2R2A, RAD51B, RAD51C, RAD51D, or other DNA repair genes) have been accrued in the first and second stage combined, then the trial will proceed with enrichment. If 3 or more subjects with those mutations have been accrued, then enrichment will again proceed as long as the response rate in that subject of subjects is ≥20%.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of adenocarcinoma of the prostate
2. Prior local therapy with prostatectomy required, with available tissue from prostatectomy specimen to send for genomic and transcriptomic testing.
3. Prior salvage or adjuvant radiation therapy is allowed but not mandated. Radiation therapy must have been completed for at least 6 months.
4. Absolute PSA ≥1 ng/ml. Prior undetectable PSA post-prostatectomy is not required.
5. PSADT ≤6 months, based upon ≥3 consecutive measurements collected in the past 12 months, at least 4 weeks apart
6. No radiographic evidence of metastatic disease by CT scan and bone scan, performed within the prior 4 weeks.
7. Serum testosterone ≥ 150 ng/dl
8. Participants must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

   * Hemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Platelet count ≥ 75 x 109/L
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) <2.5 x institutional upper limit of normal. Note: Patients with elevations in bilirubin, AST, or ALT should be thoroughly evaluated for the etiology of this abnormality prior to entry and patients with evidence of viral infection should be excluded.
   * Patients must have creatinine clearance estimated using the Cockcroft

     * Gault equation of ≥51 mL/min:

   Estimated creatinine clearance = (140-age [years]) x weight (kg) serum creatinine (mg/dL) x 72
9. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
10. Male participants and their partners, who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination [see appendix F for acceptable methods], throughout the period of taking study treatment and for 3 months after last dose of study drug to prevent pregnancy in a partner.
11. For enrichment stage of trial only (if necessary): Confirmation of a suspected/known deleterious mutation in a gene of interest (ATM, BARD1, BRCA1, BRCA2, BRIP1, CDK12, CHEK1, CHEK2, FANCL, PALB2, PPP2R2A, RAD51B, RAD51C, RAD51D, or other DNA repair genes) via CLIA certified testing.

Exclusion Criteria:

1. Prior ADT in the past 6 months. Prior ADT in context of neoadjuvant/adjuvant primary; prior ADT for biochemical recurrence is allowed, as long as no ADT has been administered in past 6 months and testosterone has recovered (>150 ng/dl). The total duration of prior ADT should not exceed 24 months.
2. Prior oral anti-androgen (e.g. bicalutamide, nilutamide, enzalutamide, apalutamide), or androgen synthesis inhibitor (e.g. abiraterone, orteronel) in the past 6 months. 5-alpha reductase inhibitor therapy (e.g. finasteride, dutasteride) is allowed, as long as subject has been stable on medication for past 6 months.
3. Prior treatment with intravenous chemotherapy.
4. Involvement in the planning and/or conduct of the study
5. Participation in another clinical study with an investigational product during the last 1 month.
6. Any previous treatment with PARP inhibitor, including olaparib
7. Resting ECG with QTc > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome
8. Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
9. Concomitant use of known strong CYP3A inducers (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for phenobarbital and 3 weeks for other agents.
10. Myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
11. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
12. Poor medical risk due to a serious, uncontrolled medical disorder, non- malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
13. Unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
14. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
15. Known hypersensitivity to olaparib or any of the excipients of the product.
16. Known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids
17. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable, for timing refer to inclusion criteria no.10)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2026-05-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine H Marshall, MD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marshall CH, Teply BA, Lu J, Oliveira L, Wang H, Mao SS, Kelly WK, Paller CJ, Markowski MC, Denmeade SR, King S, Sullivan R, Davicioni E, Proudfoot JA, Eisenberger MA, Carducci MA, Lotan TL, Antonarakis ES. Olaparib Without Androgen Deprivation for High-Risk Biochemically Recurrent Prostate Cancer Following Prostatectomy: A Nonrandomized Controlled Trial. JAMA Oncol. 2024 Oct 1;10(10):1400-1408. doi: 10.1001/jamaoncol.2024.3074. PMID 39172479

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Olaparib 300 mg BID
Started | 51
Completed | 48
Not Completed | 3
Not completed — Still being treated | 3

BASELINE CHARACTERISTICS:
Arm/Group | Olaparib 300 mg BID
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.8 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 47
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: PSA50 Response Rate to Olaparib for Patients With High-risk Biochemically-recurrent Prostate Cancer
Description: Number of participants with PSA50 response defined as at least a 50% decline in Prostate Specific Antigen (PSA) from baseline value, confirmed with a second measurement at least 4 weeks apart.
Time Frame: 6 years 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 300 mg BID
Number analyzed (Participants) | 51
Participants | 13

2. Secondary Outcome: Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: Number of participants with treatment related adverse events
Time Frame: Baseline to End of Treatment
Reporting Status: Not Posted, anticipated posting 2025-12

3. Secondary Outcome: PSA Progression-free Survival
Description: Defined as a time from initiation on olaparib therapy until PSA increase of 25%, confirmed with another measurement at least 4 weeks later.
Time Frame: 7 years
Reporting Status: Not Posted, anticipated posting 2025-12

4. Secondary Outcome: PSA Doubling From Baseline
Time Frame: 7 years
Reporting Status: Not Posted, anticipated posting 2025-12

5. Secondary Outcome: Duration of Undetectable PSA
Description: Number of patients on study with olaparib who achieves a PSA < 0.1, which is confirmed with a repeat measurement at least 12 weeks later.
Time Frame: 7 years
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: Baseline to End of Treatment approximately 6 years 2 months
Arm/Group | Olaparib 300 mg BID
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 2/51
Other Adverse Events (participants affected / at risk) | 35/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300 mg BID (N=51)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cerebrovascular Accident (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300 mg BID (N=51)
Nausea (Gastrointestinal disorders) | 28 (28)
Leukopenia (Blood and lymphatic system disorders) | 20 (20)
Fatigue (General disorders) | 35 (35)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Anorexia (Metabolism and nutrition disorders) | 10 (10)
Headache (Nervous system disorders) | 13 (13)
Dizziness (Nervous system disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 8 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (9)
Anemia (Blood and lymphatic system disorders) | 19 (19)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Dysgeusia (Nervous system disorders) | 14 (14)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Edema (General disorders) | 5 (5) — Lower Extremity
Constipation (Gastrointestinal disorders) | 5 (5)
Abdominal Pain (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 6 (6)
Pain-Back (Musculoskeletal and connective tissue disorders) | 3 (3)
Alanine Aminotransferase-Increased (Blood and lymphatic system disorders) | 5 (5)
Aspartate Aminotransferase-increased (Blood and lymphatic system disorders) | 3 (3)
Dry Mouth (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/35/NCT03047135/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT03047135/ICF_001.pdf